CLINICAL TRIAL: NCT04357834
Title: Wearable-based COVID-19 Markers for Prediction of Clinical Trajectories. The WAVE Study.
Brief Title: WAVE. Wearable-based COVID-19 Markers for Prediction of Clinical Trajectories
Acronym: WAVE
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: WAVE
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: COVID; COVID 19; SARS-CoV 2
Keywords: Smartwatch; Intensive care; Intensive care unit; Prediction; Artificial intelligence; Clinical trajectories
MeSH Terms: conditions — COVID-19 | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smartwatch group
  Interventions: Other: Equipment with smartwatch throughout hospital stay on the general ward

INTERVENTIONS:
Other: Equipment with smartwatch throughout hospital stay on the general ward — Participants with confirmed SARS-CoV-2 infection or suspicion of COVID-19 will be equipped with a smartwatch and wear the device throughout the hospital stay on the general ward.

SUMMARY:
The aim is to develop a wearable-based ICU (intensive care unit) prediction algorithm for inpatients contracted with SARS-CoV-2. Inpatients with suspicion of COVID-19 or with confirmed SARS-CoV-2 infection will be included. The participants will be equipped with a smartwatch, which gathers physiological data throughout hospitalisation.

DETAILED DESCRIPTION:
The SARS-CoV-2 pandemic puts an unprecedented burden on the healthcare system, specifically its healthcare providers and the resource demands for intensive care units (ICUs). To support effective care despite large case numbers, hospital operations urgently need improved decision support in early identification of patients at risk of an acute COVID-19 deterioration that requires ICU.

The investigators aim at developing a wearable-based ICU algorithm for inpatients contracted with SARS-CoV-2. Inpatients on the general ward with suspicion of COVID-19 or with confirmed SARS-CoV-2 infection will be included. The participant will be equipped with a smartwatch and wear the device throughout the hospital stay until the patient (1) is discharged home, (2) is transferred to the ICU, or (3) palliative care is initiated. The smartwatch collects several physiological parameters (e.g. heart rate, heart rate variability, respiration rate, oxygen saturation). The collected data will be used to develop an ICU prediction algorithm to detect patients at risk of an acute COVID-19 deterioration that requires ICU.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age >= 18 years
* Suspicion of COVID-19 or patient tested positive for SARS-CoV-2
* Hospitalisation on the general ward

Exclusion Criteria:

* Smartwatch cannot be attached around the wrist of the patient
* Direct transfer from the emergency department or external institution to ICU (i.e. no hospitalization on the general ward)
* Known allergies to components of the smartwatch
* Rejection of ICU transfer in the patient decree

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of COVID-19 or tested positive for SARS-CoV-2 that are or will be hospitalized on the general ward
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of smartwatch data in predicting ICU requirement in COVID-19 contracted inpatients quantified as the area under the receiver operator characteristics curve (AUC ROC > 0.85). | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Accuracy of the WAVE-model will be assessed using physiological data recorded by the smartwatch (Garmin vivoactive 4) during hospitalization complemented by demographic and health-related patient-information and will be analysed using applied machine learning technology for ICU prediction.

SECONDARY OUTCOMES:
Diagnostic accuracy of routine physiological data in predicting ICU requirement in COVID-19 contracted in-patients quantified as the area under the receiver operator characteristics curve (AUC ROC > 0.85). | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Accuracy of the model will be assessed using physiological data routinely recorded during hospitalization and will be analysed using applied machine learning technology for ICU prediction.
Diagnostic accuracy of predicting hospital discharge without ICU admission in COVID-19 contracted in-patients quantified as area under the receiver operator characteristics curve | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Accuracy of the model will be assessed using data on comorbidities, medication treatment during hospitalization and physiological data and will be analysed using casual machine-learning approaches
Change of heart rate from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Heart rate will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S) and using routine medical monitors.
Change of heart rate variability from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Heart rate variability will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S)
Change of skin temperature from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Skin temperature will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S)
Change of blood oxygen saturation from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Blood oxygen saturation will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S) and using routine medical monitors
Change of respiration rate from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Respiration rate will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S) and using routine medical monitors
Change of physical activity from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Physical activity will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S)
Change of stress level from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Stress level will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S)
Change of sleep pattern from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Sleep will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S)
Change of steps per day from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Steps per day will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S)
Change of systolic blood pressure from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Systolic blood pressure will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S) and using routine medical monitors
Change of diastolic blood pressure from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Diastolic blood pressure will be recorded throughout the hospitalization using a smartwatch (Garmin vivoactive 4S) and using routine medical monitors
Change of body temperature from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Body temperature will be recorded throughout the hospitalization using a routine medical thermometer
Change of oxygen partial pressure (pO2) from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Oxygen partial pressure (pO2) will be routinely assessed during the hospitalization in arterial or venous blood gas analyses
Change of CO2 partial pressure (pCO2) from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  CO2 partial pressure (pCO2) will be routinely assessed during the hospitalization in arterial or venous blood gas analyses
Change of blood pH from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Blood pH will be routinely assessed during the hospitalization in arterial or venous blood gas analyses
Change of bicarbonate from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Bicarbonate will be routinely assessed during the hospitalization in arterial or venous blood gas analyses
Change of base excess from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Base excess will be routinely assessed during the hospitalization in arterial or venous blood gas analyses
Change of oxygen flow rate from baseline (hospitalization) to ICU admission | until hospital discharge, transfer to ICU or palliative care is initiated (expected to be on average after 7-30 days)
  Oxygen flow rate will be routinely assessed during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Aristomenis Extradaktylos, Prof. MD, Study Chair — University Hospital Bern - Department of Emergency Medicine
Locations (1):
- Emergency Department, University Hospital Bern, Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Foll S, Lison A, Maritsch M, Klingberg K, Lehmann V, Zuger T, Srivastava D, Jegerlehner S, Feuerriegel S, Fleisch E, Exadaktylos A, Wortmann F. A Scalable Risk-Scoring System Based on Consumer-Grade Wearables for Inpatients With COVID-19: Statistical Analysis and Model Development. JMIR Form Res. 2022 Jun 21;6(6):e35717. doi: 10.2196/35717. PMID 35613417